CLINICAL TRIAL: NCT04867889
Title: PREGBRAIN - Magnetic Stimulation of the Brain in Depressed Pregnant Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to recruit participants
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Robert Boden, MD, ass prof, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PregBrain
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Depression; Pregnancy Related
Keywords: depression; pregnancy; transcranial magnetic stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a four week parallel randomized controlled trial, with two arms; the first following a protocol for magnetic stimulation of the brain with intermittent theta-burst stimulation (iTBS), with one session daily for four weeks, and the other the same protocol with a sham coil (both treatment arms will have 20 sessions in total). Apart from assessment of mood symptoms, treatment effects is also assessed using structural and functional magnetic resonance imaging.
  A random selection of the participating women will be invited to a sub-study and interviewed once during pregnancy as well as a second time 4-6 months postpartum. Questions will include inter alia their own description of being pregnant and depressed.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization into the study will be conducted by stratified block randomization. Randomization will be created via the RedCap system and a special assigned randomization personnel (the randomizer) not otherwise involved in the study. The randomizer has access to a set of patient identification codes to the Magpro X100 that determines if the patient will be given active or sham treatment. When a patient has been recruited to the study the rTMS operator will open next randomization envelope to achieve a patient code for the machine and will thereby be blinded to treatment allocation of the patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment iTBS (Active Comparator): Magnetic pulses of 120% of visual motor threshold applied in triplets of 50 Hz bursts, repeated at 5 Hz; 2 seconds on and 8 seconds off; 600 pulses per session; total duration of 3 min 20 s over the left DLPFC (F3), given in 20 sessions on 20 week days, one session per day.
  Interventions: Device: iTBS (intermittent theta-burst stimulation)
- Sham treatment (Sham Comparator): Sham treatment given either with a sham stimulation coil or by flipping an active coil 90 degrees.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: iTBS (intermittent theta-burst stimulation) — The iTBS treatment is a type of rTMS (repetitive transcranial magnetic stimulation), delivered with MagPro X100 stimulator and a Cool-B65 A/P coil or a conventional cool-B65 coil.
  The iTBS treatment is applied to over the dorsolateral prefrontal cortex using a standardized measuring of the anatomical landmark F3 from the 10-20 positioning system. The coil is positioned with the handle at in a 45 degree angle from the midline. The non-shielded side of the cool-B65 A/P coil is placed towards the patient, or if using the cool-B65 coil the centre of the butterfly is placed towards the patient head
  Arms: Active Treatment iTBS
Device: Sham iTBS — The sham iTBS is delivered with MagPro X100 stimulator and a Cool-B65 A/P coil.
  The coil is placed over the dorsolateral prefrontal cortex using a standardized measuring of the anatomical landmark F3 from the 10-20 positioning system. The coil is positioned with the handle at in a 45 degree angle from the midline. For all patients electrodes for transcutaneous electrical nerve stimulation (TENS) are applied and if the patient is randomized to sham treatment the shielded side of the coil will be pointing towards the patient's head and there will be a weak TENS current applied instead synchoronously. If the cool-B65 is used the coil is instead angled 90 degrees delivering the pulses into air instead
  Arms: Sham treatment

SUMMARY:
Background:

Depression during pregnancy is common, afflicting 10-20% of pregnant women. Nevertheless, many women want to avoid antidepressant treatment during pregnancy, due to the possible impact on the unborn child.

rTMS (repetitive transcranial magnetic stimulation) is a method where an electromagnetic coil is placed close to the head. Magnetic pulses will induce an electrical current in specific nerve cells, depending on how the coil is placed. Thousands of patients have been treated with rTMS to date, and the effect on depressive symptoms is well documented, although the exact mechanism of the effect is not yet fully understood. Of late, an alternative treatment regime called intermittent theta burst stimulation (iTBS) has been developed. The treatment time per session for iTBS is much shorter than standard rTMS, which will render the treatment much more clinically acceptable. rTMS in pregnancy has not been extensively studied, but seems to have good effect and few side effects.

Method:

Pregnant women (N=60) with depressive symptoms will be assessed by a psychiatrist, and women fulfilling the criteria for a moderate-severe depressive episode can be included. Participants will be randomized to either active or sham treatment. Treatment will be administered during 20 days, once daily (4 minutes per session). A psychiatrist will assess depressive symptoms before, as well as 2 and 4 weeks after, treatment start. Women randomized to the sham treatment will, after the initial blind phase, be offered active treatment, following the same protocol as above. Women who have responded to the treatment, but are not in remission after the first four weeks will be offered an additional two weeks of iTBS treatment, in accordance with clinical protocol.

Three, 6 and 12 months after the treatment is completed, all participants will be followed up via a web-based questionnaire.

Apart from assessment of mood symptoms, treatment effects is also assessed using structural and functional magnetic resonance imaging (MRI). MRI will be performed once before treatment start, and once before at the very end of the blind phase of the study (four weeks).

A random selection of the participating women will be invited to a sub-study and interviewed once during pregnancy as well as a second time 4-6 months postpartum. Questions will include inter alia their own description of being pregnant and depressed.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women over the age of 18 with a diagnosis of uni- or bipolar depression verified through a Mini International Neuropsychiatric Interview (M.I.N.I.) (44), and with unchanged medication the past month.
2. Provision of signed informed consent form

Exclusion Criteria:

1. Epilepsy, conductive ferromagnetic or other magnetic sensitive metals implanted in the head or within 30 cm of the treatment coil (examples cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents and bullet fragments), implanted device that is activated or controlled in any way by physiological signals such as pacemakers, implantable cardioverter-defibrillators (ICD's), vagus nerve stimulators, wearable cardioverter-defibrillators, implanted mediation pumps, intracardiac lines, even when removed, addiction (illicit drugs or alcohol), pre-eclampsia/eclampsia, previous preterm birth and/or treatment with any medication that could lower the threshold for seizures.
2. Any condition that seriously increases the risk of non-compliance or loss of follow-up

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Difference in MADRS-rating from baseline to day of the last treatment in the blind phase | 4 weeks
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10 item rating scale for depressive symptoms ranging from 0-60 points where a higher score indicates worse symptoms

SECONDARY OUTCOMES:
Difference in MADRS-rating from baseline to two weeks after first iTBS treatment | 4 weeks
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10 item rating scale for depressive symptoms ranging from 0-60 points where a higher score indicates worse symptoms
Duration of treatment effects of iTBS on symptoms in depression | 1 year
  Montgomery-Asberg Depression Rating Scale (MADRS) is a 10 item rating scale for depressive symptoms ranging from 0-60 points where a higher score indicates worse symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bodén, MD, ass prof, Principal Investigator — Uppsala University
Locations (1):
- Brain Stimulation Unit, Uppsala university hospital, Uppsala, Region Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol